CLINICAL TRIAL: NCT00409227
Title: Prospective Randomized Placebo Controlled Blinded Study to Evaluate the Efficacy of Alfuzosin (Alpha Blocker) on the Success Rates Following SWL.
Brief Title: Does Treatment With Alfuzosin Increase Success Rates of (SWL) Shock Wave Lithotripsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Yoram I Siegel MD, Assaf Harofeh MC
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 165/05
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Urolithiasis; Nephrolithiasis; Ureterolithiasis
Keywords: swl; lithotripsy; stone disease; urolithiasis; nephrolithiasis
MeSH Terms: conditions — Urolithiasis; Nephrolithiasis; Ureterolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): double blind placebo control
  Interventions: Drug: Alpha blocker-alfuzosin
- 2 (Placebo Comparator): placebo control blinded arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Alpha blocker-alfuzosin — P.O. alfuzosin 10 mg once a day
  Arms: 1
Drug: placebo — placebo once a day for 3 months or stone free
  Arms: 2

SUMMARY:
In latest literature more evidence is available about the positive effect of alpha blocker on stone expulsion from the ureter. Patients benefit from less pain and shortening time to stone expulsion. Our study is design to evaluate whether alfuzosin improves the stone free out come following SWL.

DETAILED DESCRIPTION:
All patients undergoing SWL are included in study. Exclusion criteria: Patient with radio-lucent stone, patients treated with calcium channel blockers, alpha blockers, steroids, patients with contraindication to alpha blocker treatment, postural hypotension patents with abnormal liver function tests.

Patient will be recruited to the study prospectively. Following signature on inform consent patients will be randomized into 2 groups. One group will be treated with alfuzosin 10mg a day and the control group with placebo. Treatment will be initiated following the lithotripsy treatment.

Parameters for investigation includes: demographic and personal data, stone size and location (obtained by CT or KUB), pain control medication and visual analogue scale assessment of pain, side effects, clinical squeals, stone free out come. Follow up evaluation will be at 1 week, 1 month, and 3 months post treatment. Success will be defined following CT evaluation at 3 months. Treatment ends at stone free achievement or at 3 months.

Endpoints:Stone free rate, time to stone free, side effect.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing shock wave lithotripsy treatment for urolithiasis.

Exclusion Criteria:

* patients with abnormal liver function, postural hypotension, alpha-blocker treatment, sensitivity to alpha-blockers, radio-lucent stone, calcium channel blocker treatment, steroids treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-12; Primary Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
use of pain control medication stone free rates | 3 months
pain visual analogue scale | 3 month
side effects | 3 months
stone free rate | 3 months
time to stone free status | 3 months
need for secondary procedures | 3 months
auxiliary procedures | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: yoram I siegel, MD, Principal Investigator — Endourology unit Urology department Assaf harofeh MC.
Locations (1):
- Endourology unit Urology department Assaf Harofeh MC, Ẕerifin, Israel